CLINICAL TRIAL: NCT02002884
Title: Prospective, Multicenter, Randomized, Double-blind, Parallel-group, Dose-response Study of Three Doses Xeomin® (incobotulinumtoxinA, NT 201) for the Treatment of Upper Limb Spasticity Alone or Combined Upper and Lower Limb Spasticity in Children and Adolescents (Age 2 - 17 Years) With Cerebral Palsy
Brief Title: Dose-response Study of Efficacy and Safety of Botulinum Toxin Type A to Treat Spasticity of the Arm(s) or of Arm(s) and Leg(s) in Cerebral Palsy
Acronym: XARA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ60201_3072_1; 2012-005496-14 (EudraCT Number)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy; Spasticity
Keywords: Upper limb spasticity; lower limb spasticity; combined upper and lower limb spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 8 Units per kg body weight incobotulinumtoxinA (Xeomin) (Experimental): 8 Units per kg body weight (maximum of 200 Units) will be injected per treated upper limb per injection cycle. Additionally, lower limb treatment may be administered, depending on clinical pattern: up to 300 Units per injection cycle. Overall maximum dose per injection cycle: 500 Units.
  Interventions: Drug: IncobotulinumtoxinA (8 Units per kg body weight)
- 6 Units per kg body weight incobotulinumtoxinA (Xeomin) (Experimental): 6 Units per kg body weight (maximum of 150 Units) will be injected per treated upper limb per injection cycle. Additionally, lower limb treatment may be administered, depending on clinical pattern: up to 225 Units per injection cycle. Overall maximum dose per injection cycle: 375 Units.
  Interventions: Drug: IncobotulinumtoxinA (6 Units per kg body weight)
- 2 Units per kg body weight incobotulinumtoxinA (Xeomin) (Experimental): 2 Units per kg body weight (maximum of 50 Units) will be injected per treated upper limb per injection cycle. Additionally, lower limb treatment may be administered, depending on clinical pattern: up to 75 Units per injection cycle. Overall maximum dose per injection cycle: 125 Units.
  Interventions: Drug: IncobotulinumtoxinA (2 Units per kg body weight)

INTERVENTIONS:
Drug: IncobotulinumtoxinA (8 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 8 Units per kg body weight incobotulinumtoxinA (Xeomin)
Drug: IncobotulinumtoxinA (6 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 6 Units per kg body weight incobotulinumtoxinA (Xeomin)
Drug: IncobotulinumtoxinA (2 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 2 Units per kg body weight incobotulinumtoxinA (Xeomin)

SUMMARY:
The purpose of this study is to determine whether injections of Botulinum toxin type A into muscles of one or both arms alone or in combination with injections into one or both legs are effective and safe in treating children/adolescents (age 2-17 years) with increased muscle tension/uncontrollable muscle stiffness (spasticity) due to cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject of 2 to 17 years of age (inclusive).
* Uni- or bilateral Cerebral Palsy (CP) with clinical need for injections with NT 201 for the treatment of upper limb (UL) spasticity at least unilaterally.
* Ashworth Scale (AS) score in the main clinical target patterns in this study:

  1. Flexed elbow: AS≥2 in elbow flexors (at least unilaterally). and/or
  2. Flexed Wrist: AS≥2 in wrist flexors (at least unilaterally).
* Clinical need according to the judgment of the investigator in one out of five treatment combinations (A-E, as shown below). AS score must be ≥2 for each target pattern chosen for injection at the Baseline Injection Visit V2.

A. UL(s) treatment only (GMFCS I-V):

A1) Unilateral treatment of UL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) for:

1. At least one of the main clinical target patterns flexed elbow (4 U/kg BW) and/or flexed wrist (2 U/kg BW).

   and
2. Additional clinical patterns in the same limb (i.e., clenched fist, thumb in palm, and/or pronated forearm) with the remaining units until maximum dose of 8 U/kg BW (maximum of 200 U) for treatment of a single UL is reached.

or

A2) Bilateral treatment of UL spasticity with equal doses of 8 U/kg BW NT 201 (maximum of 200 U) to each UL. Dose per UL must be distributed between:

1. At least one of the main clinical target patterns flexed elbow (4 U/kg BW) and/or flexed wrist (2 U/kg BW).

   and
2. Additional clinical patterns in the same limb (i.e., clenched fist, thumb in palm, and/or pronated forearm) with the remaining units until maximum dose of 8 U/kg BW (maximum of 200 U) for treatment of a single UL is reached.

B. Unilateral UL and unilateral lower limb (LL) treatment (GMFCS I-V):

B1) Unilateral treatment of UL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) for:

1. At least one of the main clinical target patterns flexed elbow (4 U/kg BW) and/or flexed wrist (2 U/kg BW).

   and
2. Additional clinical patterns in the same limb (i.e., clenched fist, thumb in palm, and/or pronated forearm) with the remaining units until maximum dose of 8 U/kg BW (maximum of 200 U) for treatment of a single UL is reached.

plus

B2) Ipsilateral unilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U). Dose to LL must be distributed to at least one of clinical target patterns pes equinus, flexed knee, adducted thigh, and extended great toe as clinically needed.

C. Unilateral UL and bilateral LL treatment (GMFCS I-III)

C1) Unilateral treatment of UL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) for:

1. At least one of the main clinical target patterns flexed elbow (4 U/kg BW) and/or flexed wrist (2 U/kg BW).

   and
2. Additional clinical patterns in the same limb (i.e., clenched fist, thumb in palm, and/or pronated forearm) with the remaining units until maximum dose of 8 U/kg BW (maximum of 200 U) for treatment of a single UL is reached.

plus

C2) Bilateral treatment of LL spasticity with 12 U/kg BW (maximum of 300 U). Dose must be distributed into at least one of clinical target patterns pes equinus, flexed knee, adducted thigh, and extended great toe, on each side. Dose distribution may vary between sides as clinically needed.

D. Unilateral UL and bilateral LL treatment (GMFCS IV and V)

D1) Unilateral treatment of UL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) for:

1. At least one of the main clinical target patterns flexed elbow (4 U/kg BW) and/or flexed wrist (2 U/kg BW).

   and
2. Additional clinical patterns in the same limb (i.e., clenched fist, thumb in palm, and/or pronated forearm) with the remaining units until maximum dose of 8 U/kg BW (maximum of 200 U) for treatment of a single UL is reached.

plus

D2) Bilateral treatment of LL spasticity with 8 U/kg BW (maximum of 200 U). Dose must be distributed into at least one of clinical target patterns pes equinus, flexed knee, adducted thigh, and extended great toe, on each side. Dose distribution may vary between sides as clinically needed.

E. Bilateral UL treatment and bilateral LL treatment (GMFCS I-III)

E1) Bilateral treatment of UL spasticity with equal doses of 8 U/kg BW NT 201 (maximum of 200 U) to each UL. Dose per UL must be distributed between

1. At least one of the main clinical target patterns flexed elbow (4 U/kg BW) and/or flexed wrist (2 U/kg BW) and
2. Additional clinical patterns in the same limb (i.e., clenched fist, thumb in palm, and/or pronated forearm) with the remaining units until maximum dose of 8 U/kg BW (maximum of 200 U) for treatment of a single UL is reached.

plus

E2) Bilateral treatment of LL spasticity with 4 U/kg BW (maximum of 100 U). Dose must be distributed into at least one of clinical target patterns pes equinus, flexed knee, adducted thigh, and extended great toe, on each side. Dose distribution may vary between sides as clinically needed.

Exclusion Criteria:

Pre-treated (non-naïve) subjects must not have received BoNT treatment within the last 14 weeks prior to Screening Visit (V1) in any indication.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 351 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (32):
- United States (6):
  - Merz Investigational Site #001286, Gulf Breeze, Florida
  - Merz Investigational Site #001284, Loxahatchee Groves, Florida
  - Merz Investigational Site #001285, Savannah, Georgia
  - Merz Investigational Site #001186, Chicago, Illinois
  - Merz Investigational Site No. #001302, Royal Oak, Michigan
  - Merz Investigational Site #001283, Columbia, Missouri
- Argentina (2):
  - Merz Investigational Site #054010, Godoy Cruz, Mendoza Province
  - Merz Investigational Site #054005, Caba
- Mexico (7):
  - Merz Investigational Site #052023, Aguascalientes
  - Merz Investigational Site #052003, Guadalajara
  - Merz Investigational Site #052024, Mexico City
  - Merz Investigational Site #052022, Mexico City
  - Merz Investigational Site #052027, Monterrey
  - Merz Investigational Site #052028, Monterrey
  - Merz Investigational Site #052026, Zapopan
- Poland (7):
  - Merz Investigational Site #048089, Bialystok
  - Merz Investigational Site #048063, Gdansk
  - Merz Investigational Site #048059, Krakow
  - Merz Investigational Site #048084, Lublin
  - Merz Investigational Site #048094, Poznan
  - Merz Investigational Site #048075, Sandomierz
  - Merz Investigational Site #048060, Wiązowna
- Russia (6):
  - Merz Investigational Site #007014, Kazan'
  - Merz Investigational Site #007015, Khabarovsk
  - Merz Investigational Site #007018, Novosibirsk
  - Merz Investigational Site #007298, Saint Petersburg
  - Merz Investigational Site #007013, Smolensk
  - Merz Investigational Site #007019, Stavropol
- Ukraine (4):
  - Merz Investigational Site #380001, Dnipropetrovsk
  - Merz Investigational Site #380005, Kharkiv
  - Merz Investigational Site #380002, Kyiv
  - Merz Investigational Site #380003, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dabrowski E, Chambers HG, Gaebler-Spira D, Banach M, Kanovsky P, Dersch H, Althaus M, Geister TL, Heinen F. IncobotulinumtoxinA Efficacy/Safety in Upper-Limb Spasticity in Pediatric Cerebral Palsy: Randomized Controlled Trial. Pediatr Neurol. 2021 Oct;123:10-20. doi: 10.1016/j.pediatrneurol.2021.05.014. Epub 2021 May 21. PMID 34339951
- [Derived] Berweck S, Banach M, Gaebler-Spira D, Chambers HG, Schroeder AS, Geister TL, Althaus M, Hanschmann A, Vacchelli M, Bonfert MV, Heinen F, Dabrowski E. Safety Profile and Lack of Immunogenicity of IncobotulinumtoxinA in Pediatric Spasticity and Sialorrhea: A Pooled Analysis. Toxins (Basel). 2022 Aug 25;14(9):585. doi: 10.3390/toxins14090585. PMID 36136523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 investigative sites in Mexico, Argentina, Russian federation, Ukraine, United States and Poland.
Pre-assignment Details: A total of 372 participants were screened, 351 participants were randomized and 350 participants were randomized and treated in the study. 331 participants completed the main period (MP) and moved to the open-label-extension period (OLEX) out of which 281 participants completed the OLEX period.
Groups:
- MP Low Dose Group: Participants in low dose group received intramuscular injections of 2 Units per kilogram (U/kg) NT 201 (maximum of 50 Units [U] in participants with greater than [>] 25 kilogram [kg] body weight [BW]) into spastic muscles of one of the upper Limb (UL) on Day 1 of MP. If the contralateral UL or one or both lower limb (LL) were also treated, participants received additional doses of NT 201. The total body dose ranged from 2 U/kg (50 U for participants with >25kg BW) to 5 U/kg (125 U for participants with >25kg BW) depending on the combination of treated limbs and the participant's Gross Motor Function Classification System (GMFCS) level.
- MP Mid Dose Group: Participants in mid dose group received intramuscular injections of 6 U/kg NT 201 (maximum of 150 U in participants with >25kg BW) into spastic muscles of one of the UL on Day 1 of MP. If the contralateral UL or one or both LL were also treated, participants received additional doses of NT 201. The total body dose ranged from 6 U/kg (150 U for participants with >25kg BW) to 15 U/kg (375 U for participants with >25kg BW) depending on the combination of treated limbs and the participant's GMFCS level.
- MP High Dose Group: Participants in high dose group received intramuscular injections of 8 U/kg NT 201 (maximum of 200 U in participants with >25kg BW) into spastic muscles of one of the UL on Day 1 of MP. If the contralateral UL or one or both LL were also treated, participants received additional doses of NT 201. The total body dose ranged from 8 U/kg (200 U for participants with >25kg BW) to 20 U/kg (500 U for participants with >25kg BW) depending on the combination of treated limbs and the participant's GMFCS level.
- OLEX (3 Injections): Participants who completed MP and qualified for further participation in the study received intramuscular injections of 8 U/kg NT 201 (maximum of 200 U in participants with >25kg BW) into spastic muscles of the UL on Day 1 of each of the three injection cycles of OLEX. If the contralateral UL or one or both LL were also treated, participants received additional doses of NT 201. The total body dose ranged from 8 U/kg (200 U for participants with >25kg BW) to 20 U/kg (500 U for participants with >25kg BW) depending on the combination of treated limbs and the participant's GMFCS level.
Period: Main Period (MP)
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Started | 87 | 88 | 176 | 0
Treated | 87 | 87 | 176 | 0
Completed | 81 | 82 | 168 | 0
Not Completed | 6 | 6 | 8 | 0
Not completed — Other | 0 | 3 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Period: Open-Label Extension Period (OLEX)
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Started | 0 | 0 | 0 | 331
Completed | 0 | 0 | 0 | 281
Not Completed | 0 | 0 | 0 | 50
Not completed — Other | 0 | 0 | 0 | 24
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants.
Groups:
- MP Low Dose Group: Participants in low dose group received intramuscular injections of 2 U/kg NT 201 (maximum of 50 U in participants with >25 kg BW) into spastic muscles of one of the UL on Day 1 of MP. If the contralateral UL or one or both LL were also treated, participants received additional doses of NT 201. The total body dose ranged from 2 U/kg (50 U for participants with >25kg BW) to 5 U/kg (125 U for participants with >25kg BW) depending on the combination of treated limbs and the participant's GMFCS level.
- Total: Total of all reporting groups
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | Total
Number analyzed (Participants) | 87 | 88 | 176 | 351
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.2 (4.70) | 7.4 (4.13) | 7.3 (4.40) | 7.3 (4.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 62 | 131
  Male | 49 | 57 | 114 | 220
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 26 | 45 | 87
  Not Hispanic or Latino | 71 | 62 | 131 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 2 | 2 | 7
  White | 81 | 75 | 160 | 316
  Other | 3 | 11 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: MP: Change From Baseline in Ashworth Scale (AS) in UL Primary Clinical Target Pattern at Week 4
Description: The AS categorizes severity of spasticity by judging resistance to passive movement. Spasticity was assessed by using the 5-point AS with:0 (no increase in tone); 1 (slight increase in tone giving a "catch" when the limb was moved in flexion or extension); 2 (more marked increase in tone, but limb easily flexed); 3 (considerable increase in tone -passive movements difficult); 4 (limb rigid in flexion or extension). Values represent least square (LS) mean differences between baseline and Week 4 resulting from Mixed Model Repeated Measurement (MMRM) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline and Week 4
Population: The full analysis set (FAS) was the subset in the safety evaluation set (SES) of the MP for whom the primary efficacy variable or co-primary efficacy variable were available. Number of participants who were evaluable for this measure at a given time period and were included in the assessment.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  High versus low: number analyzed (Participants) | 85 | 0 | 172
  High versus low | -0.93 (0.078) |  | -1.15 (0.056)
  Mid versus low: number analyzed (Participants) | 85 | 86 | 0
  Mid versus low | -0.96 (0.082) | -1.02 (0.082) |
Statistical Analysis 1: Comparison: MP Low Dose Group vs MP High Dose Group; LS-Means are from mixed model with treatment group, pooled site and pre-treatment status included as fixed factors and AS at baseline, Gross Motor Function Classification System-Extended and Revised (GMFCS-E&R) level at screening included as covariates. For MMRM visit*treatment is interaction term repeated factor; Test type: Superiority; p = 0.017, MMRM; LS Mean difference = -0.22, 95% CI 2-sided [-0.4 to -0.04]
Statistical Analysis 2: Comparison: MP Low Dose Group vs MP Mid Dose Group; LS-Means are from mixed model with treatment group, pooled site and pre-treatment status included as fixed factors and AS at baseline, GMFCS-E&R level at screening included as covariates. For MMRM visit*treatment is interaction term repeated factor; Test type: Superiority; p = 0.546, MMRM; LS-Mean difference = -0.07, 95% CI 2-sided [-0.29 to 0.15]

2. Primary Outcome: Co-primary Variable MP: Investigator's Global Impression of Change Scale (GICS) at Week 4
Description: The GICS was used to measure independently the investigator's impression of change due to treatment. The response option was a common 7-point Likert scale, that ranges from +3 (very much improved); +2 (much improved); +1 (minimally improved); 0 (no change); -1 (minimally worse); -2 (much worse); -3 (very much worse). Values represent LS mean differences between baseline and Week 4 resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Week 4
Population: The FAS was the subset in the SES of the MP for whom the primary efficacy variable or co-primary efficacy variable were available (that is, all participants who had at least an AS score in clinical pattern flexed elbow or flexed wrist at baseline [Day 1] or Investigator's GICS at Day 29 [Week 4]).
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  High versus low: number analyzed (Participants) | 87 | 0 | 176
  High versus low | 1.55 (0.083) |  | 1.64 (0.062)
  Mid versus low: number analyzed (Participants) | 87 | 87 | 0
  Mid versus low | 1.57 (0.089) | 1.44 (0.092) |
Statistical Analysis 1: Comparison: MP Low Dose Group vs MP High Dose Group; LS-Means are from analysis of covariance (ANCOVA) with treatment group, pooled site and pretreatment status included as fixed factors and maximum AS score of the two possible primary target patterns flexed elbow or flexed wrist baseline, GMFCS-E&R level at screening included as covariates; Test type: Superiority; p = 0.34, ANCOVA; LS-Mean difference = 0.09, 95% CI 2-sided [-0.1 to 0.28]
Statistical Analysis 2: Comparison: MP Low Dose Group vs MP Mid Dose Group; LS-Means are from ANCOVA with treatment group, pooled site and pre-treatment status included as fixed factors and maximum AS score of the two possible primary target patterns flexed elbow or flexed wrist baseline, GMFCS-E&R level at screening included as covariates; Test type: Superiority; p = 0.297, ANCOVA; LS-Mean difference = -0.12, 95% CI 2-sided [-0.36 to 0.11]

3. Secondary Outcome: MP: Change From Baseline in AS Score of the Other Treated UL Main Clinical Target Pattern at Week 4
Description: The AS categorizes the severity of spasticity by judging resistance to passive movement. Spasticity was assessed by 5-point scale at visits, where: 0 (no increase in tone); 1(slight increase in tone giving a "catch" when the limb was moved in flexion or extension); 2(more marked increase in tone, but limb easily flexed); 3(considerable increase in tone - passive movements difficult); 4(limb rigid in flexion or extension). Values represent LS mean differences between baseline and Week 4 resulting from MMRM models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline and Week 4
Population: The FAS was the subset in the SES of the MP for whom the primary efficacy variable or co-primary efficacy variable were available. Number of participants who were evaluable for this measure at a given time period and were included in the assessment.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  High versus low: number analyzed (Participants) | 67 | 0 | 143
  High versus low | -1.03 (0.083) |  | -1.13 (0.061)
  Mid versus low: number analyzed (Participants) | 67 | 69 | 0
  Mid versus low | -1.08 (0.087) | -1.22 (0.090) |

4. Secondary Outcome: MP: Change From Baseline in AS Score in UL Treated Clenched Fist With Flexed Wrist at Week 4
Description: as for outcome 3
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  High versus low: number analyzed (Participants) | 18 | 0 | 45
  High versus low | -0.53 (0.212) |  | -1.00 (0.133)
  Mid versus low: number analyzed (Participants) | 18 | 20 | 0
  Mid versus low | -0.070 (0.202) | -1.04 (0.176) |

5. Secondary Outcome: MP: Change From Baseline in AS Score for Each Treated Clinical Pattern of the UL at Week 4
Description: as for outcome 3
Time Frame: Baseline up to Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  Flexed elbow: High versus Low: number analyzed (Participants) | 83 | 0 | 166
  Flexed elbow: High versus Low | -0.99 (0.076) |  | -1.18 (0.056)
  Flexed elbow: Mid versus Low: number analyzed (Participants) | 83 | 82 | 0
  Flexed elbow: Mid versus Low | -1.01 (0.081) | -1.17 (0.082) |
  Flexed wrist: High versus Low: number analyzed (Participants) | 69 | 0 | 149
  Flexed wrist: High versus Low | -0.96 (0.085) |  | -1.08 (0.061)
  Flexed wrist: Mid versus Low: number analyzed (Participants) | 69 | 73 | 0
  Flexed wrist: Mid versus Low | -1.01 (0.087) | -1.05 (0.087) |
  Clenched fist: High versus Low: number analyzed (Participants) | 34 | 0 | 64
  Clenched fist: High versus Low | -0.64 (0.136) |  | -1.09 (0.096)
  Clenched fist: Mid versus Low: number analyzed (Participants) | 34 | 30 | 0
  Clenched fist: Mid versus Low | -0.58 (0.145) | -0.87 (0.141) |
  Thumb in palm: High versus Low: number analyzed (Participants) | 49 | 0 | 98
  Thumb in palm: High versus Low | -0.88 (0.116) |  | -1.11 (0.083)
  Thumb in palm: Mid versus Low: number analyzed (Participants) | 49 | 44 | 0
  Thumb in palm: Mid versus Low | -0.93 (0.131) | -1.14 (0.123) |
  Pronated forearm: High versus Low: number analyzed (Participants) | 72 | 0 | 150
  Pronated forearm: High versus Low | -0.88 (0.080) |  | -1.02 (0.058)
  Pronated forearm: Mid versus Low: number analyzed (Participants) | 72 | 73 | 0
  Pronated forearm: Mid versus Low | -0.87 (0.086) | -0.94 (0.088) |

6. Secondary Outcome: MP: Change From Baseline in Scores of Pain Intensity (From Participants) and Pain Frequency (From Parent/Caregiver) Assessed With 'Questionnaire on Pain Caused by Spasticity (QPS)'
Description: Pain intensity (from participants) and pain frequency (from parent/caregiver) to be assessed with QPS. The QPS Total Score for pain intensity ranges from 0 ('No Hurt') to 10 ('Hurt Worst'). The QPS Total Score for the observed pain frequency ranges from 0 (Never) to 4 (Always). Values represent LS mean differences between baseline and Week 4 resulting from MMRM models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison. P/C = Parent/Caregiver.
Time Frame: Baseline, Weeks 4, 8, and 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  UL, Participant, Week 4 High versus low: number analyzed (Participants) | 30 | 0 | 52
  UL, Participant, Week 4 High versus low | -0.42 (0.217) |  | -0.75 (0.199)
  UL, Participant, Week 4 Mid versus low: number analyzed (Participants) | 30 | 34 | 0
  UL, Participant, Week 4 Mid versus low | -0.39 (0.256) | -0.67 (0.289) |
  UL, Participant, Week 8 High versus low: number analyzed (Participants) | 29 | 0 | 52
  UL, Participant, Week 8 High versus low | -0.52 (0.206) |  | -0.64 (0.188)
  UL, Participant, Week 8 Mid versus low: number analyzed (Participants) | 29 | 34 | 0
  UL, Participant, Week 8 Mid versus low | -0.63 (0.259) | -0.55 (0.290) |
  UL, Participant, Week 14 High versus low: number analyzed (Participants) | 27 | 0 | 52
  UL, Participant, Week 14 High versus low | -0.56 (0.217) |  | -0.59 (0.202)
  UL, Participant, Week 14 Mid versus low: number analyzed (Participants) | 27 | 32 | 0
  UL, Participant, Week 14 Mid versus low | -0.66 (0.327) | -0.59 (0.361) |
  UL, P/C, Week 4 High versus low: number analyzed (Participants) | 64 | 0 | 133
  UL, P/C, Week 4 High versus low | -0.46 (0.102) |  | -0.44 (0.076)
  UL, P/C, Week 4 Mid versus low: number analyzed (Participants) | 64 | 65 | 0
  UL, P/C, Week 4 Mid versus low | -0.43 (0.106) | -0.28 (0.115) |
  UL, P/C, Week 8 High versus low: number analyzed (Participants) | 67 | 0 | 138
  UL, P/C, Week 8 High versus low | -0.40 (0.095) |  | -0.44 (0.070)
  UL, P/C, Week 8 Mid versus low: number analyzed (Participants) | 67 | 66 | 0
  UL, P/C, Week 8 Mid versus low | -0.43 (0.100) | -0.34 (0.109) |
  UL, P/C, Week 14 High versus Low: number analyzed (Participants) | 58 | 0 | 137
  UL, P/C, Week 14 High versus Low | -0.23 (0.105) |  | -0.24 (0.071)
  UL, P/C, Week 14 Mid versus Low: number analyzed (Participants) | 58 | 61 | 0
  UL, P/C, Week 14 Mid versus Low | -0.31 (0.100) | -0.25 (0.107) |
  LL, Participant, Week 4 High versus Low: number analyzed (Participants) | 24 | 0 | 43
  LL, Participant, Week 4 High versus Low | -0.74 (0.282) |  | -0.62 (0.250)
  LL, Participant, Week 4 Mid versus Low: number analyzed (Participants) | 24 | 29 | 0
  LL, Participant, Week 4 Mid versus Low | -0.46 (0.305) | -0.55 (0.321) |
  LL, Participant, Week 8 High versus Low: number analyzed (Participants) | 25 | 0 | 44
  LL, Participant, Week 8 High versus Low | -1.04 (0.241) |  | -0.69 (0.218)
  LL, Participant, Week 8 Mid versus Low: number analyzed (Participants) | 25 | 28 | 0
  LL, Participant, Week 8 Mid versus Low | -0.90 (0.261) | -0.81 (0.284) |
  LL, Participant, Week 14 High versus Low: number analyzed (Participants) | 23 | 0 | 43
  LL, Participant, Week 14 High versus Low | -0.71 (0.275) |  | -0.57 (0.245)
  LL, Participant, Week 14 Mid versus Low: number analyzed (Participants) | 23 | 28 | 0
  LL, Participant, Week 14 Mid versus Low | -0.67 (0.315) | -0.63 (0.335) |
  LL, P/C, Week 4 High versus Low: number analyzed (Participants) | 56 | 0 | 110
  LL, P/C, Week 4 High versus Low | -0.50 (0.105) |  | -0.52 (0.077)
  LL, P/C, Week 4 Mid versus Low: number analyzed (Participants) | 56 | 54 | 0
  LL, P/C, Week 4 Mid versus Low | -0.46 (0.103) | -0.42 (0.111) |
  LL, P/C, Week 8 High versus Low: number analyzed (Participants) | 59 | 0 | 113
  LL, P/C, Week 8 High versus Low | -0.56 (0.098) |  | -0.51 (0.074)
  LL, P/C, Week 8 Mid versus Low: number analyzed (Participants) | 59 | 54 | 0
  LL, P/C, Week 8 Mid versus Low | -0.52 (0.102) | -0.36 (0.111) |
  LL, P/C, Week 14 High versus Low: number analyzed (Participants) | 53 | 0 | 110
  LL, P/C, Week 14 High versus Low | -0.33 (0.108) |  | -0.32 (0.078)
  LL, P/C, Week 14 Mid versus Low: number analyzed (Participants) | 53 | 53 | 0
  LL, P/C, Week 14 Mid versus Low | -0.37 (0.086) | -0.31 (0.090) |

7. Secondary Outcome: MP: Child's/Adolescent's, and Parent's/Caregiver's GICS in UL at Week 4
Description: The GICS was used to measure independently the child's/adolescent's, and parent's or caregiver's impression of change due to treatment. The response option was a common 7-point Likert scale, that ranges from: +3(very much improved); +2(much improved); +1(minimally improved); 0(no change); -1(minimally worse); -2(much worse); -3(very much worse). Values represent LS mean differences between baseline and Week 4 resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group
Number analyzed (Participants) | 87 | 87 | 176
Unit on a scale
  Participant: High versus Low: number analyzed (Participants) | 31 | 0 | 55
  Participant: High versus Low | 1.51 (0.153) |  | 1.63 (0.139)
  Participant: Mid versus Low: number analyzed (Participants) | 31 | 38 | 0
  Participant: Mid versus Low | 1.53 (0.180) | 1.48 (0.190) |
  Parent/Caregiver: High versus Low: number analyzed (Participants) | 87 | 0 | 176
  Parent/Caregiver: High versus Low | 1.41 (0.087) |  | 1.60 (0.065)
  Parent/Caregiver: Mid versus Low: number analyzed (Participants) | 87 | 87 | 0
  Parent/Caregiver: Mid versus Low | 1.36 (0.094) | 1.29 (0.097) |

8. Secondary Outcome: Number of Participants With Occurrence of Treatment Emergent Adverse Events (TEAEs) Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: The SES was the subset of all participants treated in the MP and OLEX with study medication at least once. Number of participants who were evaluable for this measure at a given time period and were included in the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall | 21 | 13 | 42 | 114
  First injection cycle (MP): number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP) | 21 | 13 | 42 |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX) |  |  |  | 64
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX) |  |  |  | 42
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX) |  |  |  | 48

9. Secondary Outcome: Number of Participants With Occurrence of TEAEs of Special Interest (TEAESIs) Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall | 1 | 1 | 1 | 5
  First injection cycle (MP): number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP) | 1 | 1 | 1 |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX) |  |  |  | 2
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX) |  |  |  | 3
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX) |  |  |  | 1

10. Secondary Outcome: Number of Participants With Occurrence of Serious TEAEs (TESAEs) Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: The SES were the subset of all participants treated in the MP and OLEX with study medication at least once. Number of participants who were evaluable for this measure at a given time period and were included in the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall | 2 | 1 | 2 | 16
  First injection cycle (MP): number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP) | 2 | 1 | 2 |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX) |  |  |  | 7
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX) |  |  |  | 9
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX) |  |  |  | 3

11. Secondary Outcome: Number of Participants With Occurrence of TEAEs Related to Treatment Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: The SES was the subset of all participants treated in MP and OLEX with study medication at least once. Number of participants who were evaluable for this measure at a given time period and were included in the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall | 0 | 0 | 3 | 5
  First injection cycle (MP): number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP) | 0 | 0 | 3 |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX) |  |  |  | 2
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX) |  |  |  | 2
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX) |  |  |  | 1

12. Secondary Outcome: Number of Participants With Occurrence of TEAEs by Worst Intensity Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall: Mild | 15 | 10 | 33 | 62
  Overall: Moderate | 6 | 2 | 7 | 44
  Overall: Severe | 0 | 1 | 2 | 8
  First injection cycle (MP): Mild: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Mild | 15 | 10 | 33 |
  First injection cycle (MP): Moderate: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Moderate | 6 | 2 | 7 |
  First injection cycle (MP): Severe: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Severe | 0 | 1 | 2 |
  Second injection cycle (OLEX): Mild: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Mild |  |  |  | 43
  Second injection cycle (OLEX): Moderate: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Moderate |  |  |  | 18
  Second injection cycle (OLEX): Severe: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Severe |  |  |  | 3
  Third injection cycle (OLEX): Mild: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Mild |  |  |  | 23
  Third injection cycle (OLEX): Moderate: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Moderate |  |  |  | 15
  Third injection cycle (OLEX): Severe: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Severe |  |  |  | 4
  Fourth injection cycle (OLEX): Mild: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Mild |  |  |  | 28
  Fourth injection cycle (OLEX): Moderate: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Moderate |  |  |  | 19
  Fourth injection cycle (OLEX): Severe: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Severe |  |  |  | 1

13. Secondary Outcome: Number of Participants With Occurrence of TEAEs by Worst Causal Relationship Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall: Related | 0 | 0 | 3 | 5
  Overall: Not related | 21 | 13 | 39 | 109
  First injection cycle (MP): Related: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Related | 0 | 0 | 3 |
  First injection cycle (MP): Not related: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Not related | 21 | 13 | 39 |
  Second injection cycle (OLEX): Related: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Related |  |  |  | 2
  Second injection cycle (OLEX): Not related: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Not related |  |  |  | 62
  Third injection cycle (OLEX): Related: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Related |  |  |  | 2
  Third injection cycle (OLEX): Not related: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Not related |  |  |  | 40
  Fourth injection cycle (OLEX): Related: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Related |  |  |  | 1
  Fourth injection cycle (OLEX): Not related: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Not related |  |  |  | 47

14. Secondary Outcome: Number of Participants With Occurrence of TEAEs by Final Outcome Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall: Resolved | 18 | 10 | 39 | 96
  Overall: Resolved with sequelae | 1 | 0 | 0 | 1
  Overall: Resolving | 0 | 2 | 1 | 7
  Overall: Not resolved | 2 | 1 | 1 | 8
  Overall: Unknown | 0 | 0 | 1 | 2
  Overall: Fatal | 0 | 0 | 0 | 0
  First injection cycle (MP): Resolved: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Resolved | 18 | 10 | 39 |
  First injection cycle (MP): Resolved with sequelae: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Resolved with sequelae | 1 | 0 | 0 |
  First injection cycle (MP): Resolving: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Resolving | 0 | 2 | 1 |
  First injection cycle (MP): Not resolved: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Not resolved | 2 | 1 | 1 |
  First injection cycle (MP): Unknown: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Unknown | 0 | 0 | 1 |
  First injection cycle (MP): Fatal: number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP): Fatal | 0 | 0 | 0 |
  Second injection cycle (OLEX): Resolved: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Resolved |  |  |  | 57
  Secondinjection cycle(OLEX):Resolved with sequelae: number analyzed (Participants) | 0 | 0 | 0 | 331
  Secondinjection cycle(OLEX):Resolved with sequelae |  |  |  | 0
  Second injection cycle (OLEX): Resolving: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Resolving |  |  |  | 3
  Second injection cycle (OLEX): Not resolved: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Not resolved |  |  |  | 4
  Second injection cycle (OLEX): Unknown: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Unknown |  |  |  | 0
  Second injection cycle (OLEX): Fatal: number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX): Fatal |  |  |  | 0
  Third injection cycle (OLEX): Resolved: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Resolved |  |  |  | 37
  Third injection cycle(OLEX):Resolved with sequelae: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle(OLEX):Resolved with sequelae |  |  |  | 0
  Third injection cycle (OLEX): Resolving: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Resolving |  |  |  | 0
  Third injection cycle (OLEX): Not resolved: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Not resolved |  |  |  | 4
  Third injection cycle (OLEX): Unknown: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Unknown |  |  |  | 1
  Third injection cycle (OLEX): Fatal: number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX): Fatal |  |  |  | 0
  Fourth injection cycle (OLEX): Resolved: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Resolved |  |  |  | 39
  Fourthinjection cycle(OLEX):Resolved with sequelae: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourthinjection cycle(OLEX):Resolved with sequelae |  |  |  | 1
  Fourth injection cycle (OLEX): Resolving: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Resolving |  |  |  | 4
  Fourth injection cycle (OLEX): Not resolved: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Not resolved |  |  |  | 2
  Fourth injection cycle (OLEX): Unknown: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Unknown |  |  |  | 2
  Fourth injection cycle (OLEX): Fatal: number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX): Fatal |  |  |  | 0

15. Secondary Outcome: Number of Participants With Occurrence of TEAEs Leading to Discontinuation Overall and Per Treatment Cycle
Time Frame: Baseline up to Week 66
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
Number analyzed (Participants) | 87 | 87 | 176 | 331
Participants
  Overall | 0 | 1 | 1 | 5
  First injection cycle (MP): number analyzed (Participants) | 87 | 87 | 176 | 0
  First injection cycle (MP) | 0 | 1 | 1 |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Second injection cycle (OLEX) |  |  |  | 3
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Third injection cycle (OLEX) |  |  |  | 2
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 331
  Fourth injection cycle (OLEX) |  |  |  | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 66
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | MP Low Dose Group | MP Mid Dose Group | MP High Dose Group | OLEX (3 Injections)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/87 | 0/176 | 0/331
Serious Adverse Events (participants affected / at risk) | 2/87 | 1/87 | 2/176 | 16/331
Other Adverse Events (participants affected / at risk) | 5/87 | 3/87 | 6/176 | 18/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP Low Dose Group (N=87) | MP Mid Dose Group (N=87) | MP High Dose Group (N=176) | OLEX (3 Injections) (N=331)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CSF shunt operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electroencephalogram (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP Low Dose Group (N=87) | MP Mid Dose Group (N=87) | MP High Dose Group (N=176) | OLEX (3 Injections) (N=331)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (5) | 6 (6) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2016-04-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT02002884/Prot_001.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02002884/SAP_000.pdf